CLINICAL TRIAL: NCT06264440
Title: A Phase 1, Open-Label, Crossover Study to Assess the Potential for Gastric pH-Dependent Drug-Drug Interactions of BIIB122 With a Proton Pump Inhibitor in Healthy Participants
Brief Title: A Study to Assess the Potential for Gastric-pH Dependent Drug-Drug Interactions of BIIB122 With a Proton Pump Inhibitor in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 283HV104
Record Dates: First submitted 2024-02-09; First posted 2024-02-20 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — DNL151; Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Period 1 (Experimental): Participants will receive a single oral dose of BIIB122, while fasting, followed by a washout period.
  Interventions: Drug: BIIB122
- Period 2 (Experimental): Participants will receive PPI pretreatment (rabeprazole) once daily (QD), followed by a single oral dose of BIIB122 while fasting, followed by a washout period.
  Interventions: Drug: BIIB122; Drug: Rabeprazole
- Period 3 (Experimental): Participants will receive PPI pretreatment (rabeprazole) QD, followed by a single oral dose of BIIB122 while fed, followed by a washout period.
  Interventions: Drug: BIIB122; Drug: Rabeprazole

INTERVENTIONS:
Drug: BIIB122 — Administered as specified in the treatment arm.
  Other Names: DNL151
Drug: Rabeprazole — Administered as specified in the treatment arm.
  Arms: Period 2; Period 3

SUMMARY:
The primary objective of the study is to evaluate the effects of a proton pump inhibitor (PPI) [rabeprazole] on BIIB122 pharmacokinetics (PK) after a single dose in healthy participants. The secondary objective of the study is to evaluate the safety and tolerability of BIIB122, with and without a PPI (rabeprazole), after a single dose in healthy participants.

ELIGIBILITY:
Key Inclusion Criteria:

1. Body mass index between 18 and 30 kilograms per square meter (kg/^m2), inclusive.

3. Negative polymerase chain reaction test result for severe acute respiratory syndrome coronavirus (SARS-CoV-2) at Check-in.

4. For participants ≥ 55 years of age, ongoing conditions must be considered by the Investigator to be stable and adequately controlled by allowed concomitant medications.

Key Exclusion Criteria:

1. Plans to undergo elective procedures or surgeries at any time after signing the Informed Consent Form (ICF) through the follow-up visit.
2. Any condition affecting study treatment absorption.
3. History of gastrointestinal surgery, gastroesophageal reflux disease, or other clinically significant and active gastrointestinal condition per the Investigator's discretion.
4. Clinically significant acute gastrointestinal symptoms within 30 days prior to study Check-in (Day -1).
5. Chronic, recurrent, or serious infection, as determined by the Investigator, within 90 days prior to Screening or between Screening and Day -1.
6. For participants < 55 years of age: Use of any prescription medication (excluding oral contraceptives and hormone replacement therapy), OTC oral medications including proton pump inhibitors (PPI), histamine H2-receptor antagonists (H2 blockers), and antacids (excluding acetaminophen and aspirin ≤ 100 mg daily), or nutraceuticals including vitamins/mineral supplements/herbal medicines within 28 days prior to Day -1 and throughout the study.
7. For participants ≥ 55 years of age: Up to 5 medications are allowed if they are taken at a stable dose level and regimen.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2024-02-12 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Concentration (Cmax) of BIIB122 | Up to Day 55
Area Under the Concentration-Time Curve From Time Zero to Time of the Last Measurable Concentration (AUClast) of BIIB122 | Up to Day 55
Area Under the Concentration-Time Curve From Time Zero to Infinity (AUCinf) of BIIB122 | Up to Day 55

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Day 55

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- PPD Development, LP, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/